CLINICAL TRIAL: NCT04366999
Title: Effectiveness of Bariatric Surgery for Nonalcoholic Fatty Liver Diseases/Nonalcoholic Steatohepatitis With Fibrosis : A Prospective, Multicentric Cohort Study
Brief Title: Effectiveness of Bariatric Surgery for NAFLD/NASH
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Beijing Hospital (only for Base-NAFLD) (Unknown); Beijing Shijitan Hospital, Capital Medical University Beijing Hospital (only for Base-NAFLD) (Unknown); Shanghai Jiao Tong University affiliated Sixth People's Hospital Beijing Hospital (only for Base-NAFLD) (Unknown); Huashan Hospital, Fudan University Beijing Hospital (only for Base-NAFLD) (Unknown); Beijing Chao Yang Hospital (Other); Capital Medical University (Other); The First Hospital of Kunming (Unknown); Bishan Hospital of Chongqiang Medical University (Unknown); The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Director of general surgery, principal investigator, Beijing Friendship Hospital
Other Study IDs: Base-NAFLD/NASH
Record Dates: First submitted 2020-04-21; First posted 2020-04-29 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Bariatric Surgery Candidate; NAFLD; NASH With Fibrosis
Keywords: Bariatric surgery; NAFLD; NASH; Fibrosis; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Paired liver biopsy: Intraoperative, at least 1-year after surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SG: In this group, the bariatric procedure is sleeve gastrectomy (SG), all operations follow the same standard operating procedure.
  Interventions: Procedure: SG
- RYGB: In this group, the bariatric procedure is Roux-en-Y gastric bypass (RYGB), all operations follow the same standard operating procedure.
  Interventions: Procedure: RYGB
- OAGB: In this group, the bariatric procedure is one anastomosis gastric bypass(OAGB), all operations follow the same standard operating procedure.
  Interventions: Procedure: OAGB

INTERVENTIONS:
Procedure: SG — SG involved a vertical gastric resection beginning 4-6 cm from the pylorus and ending 1-2 cm from the His angle, using linear staplers with the guidance of a 36 French intragastric bougie.
  Groups: SG
Procedure: RYGB — RYGB entails the creation of a 15-30 mL (approximate) gastric pouch, a 150 cm Roux limb, and a 50 cm biliopancreatic limb.
  Groups: RYGB
Procedure: OAGB — OAGB entails the creation of a long gastric tube by beginning 2 cm below the angular incisure starting from the lesser curvature side and then divided vertically upward by linear cutting staplers as calibrated with a 36 French bougie, followed by the creation of a single gastrojejunal anastomosis with an afferent biliopancreatic limb of 200 cm.
  Groups: OAGB

SUMMARY:
This is a prospective, multicenter cohort study, which subjects were obese patients requiring bariatric surgery.

This study aims to explore the the effectiveness of bariatric surgery for NAFLD/NASH with fribrosis, to explore the differences in the effectiveness among sleeve gastrostomy [SG], Roux-en-Y gastric bypass [RYGB], or one anastomosis gastric bypass [OAGB], and to explore the independent effectiveness of bariatric surgery in histological remission of NAFLD/NASH.

The first stage of the cohort was started in 2020, named Base-NAFLD; In May 2024, based on Base-NAFLD, we plan to continue established a secondary cohort, named Base-NASH.

ELIGIBILITY:
Inclusion Criteria:

[For Base-NAFLD]

1. Age between 16 and 65 years (all sexes).
2. Diagnosed with obesity according to the World Health Organization criteria for obesity in Asian populations and scheduled for a primary bariatric surgery at the participating centres.
3. Diagnosed with hepatic steatosis preoperatively by radiologic (including ultrasonography, magnetic resonance imaging [MRI]-derived proton density fat fraction [PDFF]) or pathologic(intraoperative hepatic pathology) examinations.

[For Base-NASH]

1. Age between 16 and 65 years (all sexes).
2. Diagnosed with obesity according to the World Health Organization criteria for obesity in Asian populations and scheduled for a primary bariatric surgery at the participating centres.
3. Histologically confirmed NASH with fibrosis:

NAFLD activity score(NAS) ≥4 with at least 1 in each single item and NASH-CRN fibrosis stage ≥F1

Exclusion Criteria:

* any patient who had previously been submitted to any type of bariatric surgery;
* history of excessive drinking: in the past 12 months, the male equivalent of alcohol consumption more than 30g/d, and the female more than 20g/d;
* history of taking amiodarone, methotrexate, tamoxifen, glucocorticoids, etc.；
* history of specific diseases: Gene type 3 hepatitis C virus (HCV) infection, hepatolenticular degeneration, autoimmune hepatitis, total parenteral nutrition, lack of beta lipoproteinemia, congenital lipid atrophy, celiac disease which causing fatty liver, etc.;
* previous major gastrointestinal surgery；
* diagnosed or suspected malignancy；
* poorly controlled significant medical or psychiatric disorders；
* disorders such as a medical history of major pathology;
* can not be able to understand and willing to participate in this registry with signature.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise male and non-pregnant female patients, aged 16-65years both inclusive, with morbid obesity.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the remisson rate of NAFLD (for Base-NAFLD cohort) | 1 years after surgery
  Percentage of liver fat content <5% of abdominal magnetic resonance imaging(MRI) at 1 year after surgery.
  Visit : Post-op 12 months (±30 Days)
Histological remission of NASH without worsening of fibrosis (for Base-NASH cohort) | 1 years after surgery
  *NASH resolution was defined as presence of a CRN inflammation score of 0 or 1 and no hepatocyte ballooning (score of 0).
  **Worsening of fibrosis was defined as an increase of one stage or more on the NASH-CRN fibrosis score at 1-year follow-up.

SECONDARY OUTCOMES:
the rate of fibrosis improvement without NASH worsening | 1 year after surgery
  NASH worsening, was defined as an increase of ≥1 point in either the lobular inflammation score or the hepatocyte ballooning score.
changes in NASH and liver fbrosis biopsy fndings | 1 year after surgery
  2．including the NAS (NAFLD activity score) and SAF scores (steatosis [S], activity [A], and fbrosis [F]) .
changes in body weight | 3 months, 6 months, and 1 year after surgery
  1. percent excess weight loss (%EWL): %EWL=([initial weight] - [postoperative weight])/([initial weight] - [ideal weight]) (idealweight is defned as a body mass index [BMI] of 25 kg/m2 at each follow-up point)
  2. percentage of total weight loss (%TWL): %TWL=([initial weight] - [postoperative weight])/([initial weight])×100
resolution of obesity-related comorbidities | 1 year after surgery
  4．blood glucose levels, lipid levels, and liver enzyme levels.
incidence of adverse health events | 1 year after surgery
  Including but not limited to bleeding, ulcer, intestinal obstruction etc.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, M.D.;Ph.D., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wei L, Li M, Zeng N, Liu Y, Bai R, Zhang N, Song J, Zhang P, Yao Q, Yang Z, Zhao X, Zhang Y, Zhang P, Zhang Z. Bariatric surgery for non-alcoholic fatty liver disease in individuals with obesity (Base-NAFLD): protocol of a prospective multicenter observational follow-up study. BMC Surg. 2021 Jun 24;21(1):298. doi: 10.1186/s12893-021-01296-y. PMID 34167531